CLINICAL TRIAL: NCT01315626
Title: Identification of Patients With a Diagnosis of Bronchiectasis: Evaluation of an Educational Intervention
Brief Title: Bronchiectasis: Evaluation of an Educational Intervention
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor did not move forward with study
Sponsor: Hill-Rom (Industry)
Responsible Party: Sponsor
Other Study IDs: CR-2010-04
Record Dates: First submitted 2010-12-20; First posted 2011-03-15 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2011-03

CONDITIONS: Bronchiectasis
Keywords: Bronchiectasis; pulmonary exacerbations; pulmonary infections
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Immediately preceding intervention: 3 months immediately before the education event. Charts of patients with a primary respiratory complaint will be reviewed so evaluate if they 1) have experienced 3 or more suppurative respiratory infections and 2) have required 3 or more courses of antibiotic therapy for respiratory infection over the period of one year. 4) Whether or not they underwent a HRCT, and if so, and 5) Were the patients diagnosed with BE.
- 3 months after educational event: 3 months immediately after the education event. An active assessment will be preformed as per the proposed diagnostic algorithm (attachment B) Patients that meet all criteria in the algorithm are considered at risk for bronchiectasis and based on these criteria, physicians will be encouraged to order HRCT, and the number/ proportion of patients identified with BE will be noted and compared to the other time periods.
  Interventions: Other: Primary Care Educational event
- Seasonal prior year: As respiratory illnesses are commonly seasonal, an assessment of rate of Bronchiectasis diagnosis during the months of Period 2 in the year prior to the educational intervention will also be assessed as described in Period 1
  Interventions: Other: Primary Care Educational event

INTERVENTIONS:
Other: Primary Care Educational event — The purpose of this study is to assess the accuracy of primary care physicians in diagnosing BE and evaluate the impact of an educational intervention targeting those primary care physicians and providing instruction in the recognition and treatment of BE. The hope is that a better understanding of the disease will result in more accurate diagnoses and ultimately in more appropriate care for these patients. In addition to better care for patients, earlier recognition of bronchiectasis may result in a decrease in health care costs.
  Groups: 3 months after educational event; Seasonal prior year

SUMMARY:
A study of an educational intervention of primary care practice physicians to assist in the identification of patients who have Bronchiectasis and to assess the effectiveness of the specific didactic educational intervention targeting primary care physicians in the recognition of Bronchiectasis.

DETAILED DESCRIPTION:
A pilot study will be conducted for the purpose of evaluating an educational intervention (Description in Appendix A). As part of the educational intervention, primary care physician(s) will be trained in the use of an algorithm to guide assessment of patients seen with a respiratory chief complaint, and who have not previously been identified as having a diagnosis of BE. We propose an evaluation of three primary care practice(s) to compare the number of patients identified in three three-month periods as having a diagnosis of BE.

The evaluation periods will be as follows: Period 1) the three-month period immediately following the intervention, Period 2) the three-month period immediately preceding the intervention, Period 3) the three month period starting one year prior to the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Respiratory is the chief complaint
2. Patient > 35 years of age
3. Seen in practice for > 12 months

Exclusion Criteria:

1) Prior diagnosis with bronchiectasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present, or who have been seen in the above time periods, to the participating primary care physician with the following inclusion / exclusion criteria will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2011-02 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
Number / Percent of BE patients | 18 months
  The primary outcome for this study will be the number/proportion of patients that meet entrance criteria that are subsequently diagnosed with bronchiectasis.

SECONDARY OUTCOMES:
HRCT patients | 18 months
  Secondary outcomes are the number/proportion of those subjects that undergo HRCT, and the number/proportion of subjects that are then identified as having Bronchiectasis.

CONTACTS AND LOCATIONS:
Locations (1):
- Howard Rupard, MD Primary Care Practice, Shelbyville, Tennessee, United States